CLINICAL TRIAL: NCT04360824
Title: COVID-19-associated Coagulopathy: Safety and Efficacy of Prophylactic Anticoagulation Therapy in Hospitalized Adults With COVID-19
Brief Title: Covid-19 Associated Coagulopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Usha Perepu, Sponser Investigator, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202004235
Record Dates: First submitted 2020-04-13; First posted 2020-04-24 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-01

CONDITIONS: COVID 19 Associated Coagulopathy

STUDY DESIGN:
Intervention Model Description: This is a multi-center, randomized, open-label study comparing standard prophylactic dose enoxaparin (40 mg SC daily or 30 or 40 mg SC twice daily if BMI ≥30kg/m2; standard of care arm) versus intermediate-dose enoxaparin (1 mg/kg SC daily or 0.5 mg/kg SC twice daily if BMI≥30kg/m2; intervention arm) in hospitalized patients with laboratory-confirmed SARS-CoV-2 infection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): 1) Patients randomized to the standard of care arm will receive standard prophylactic dose enoxaparin (40 mg subcutaneously daily if BMI <30kg/m2 and 30 mg subcutaneously twice daily or 40 mg subcutaneously twice daily if BMI ≥ 30kg/m2).
  Interventions: Drug: Standard of Care thromboprophylaxis
- Interventional (Other): 2) Patients randomized to the intervention arm will receive intermediate-dose enoxaparin (1 mg/kg Subcutaneously daily if BMI<30 kg/m2 or 0.5 mg/kg Subcutaneously twice daily if BMI ≥ 30kg/m2).
  Interventions: Drug: Intermediate dose thromboprophylaxis

INTERVENTIONS:
Drug: Intermediate dose thromboprophylaxis — 2) Patients randomized to the intervention arm will receive intermediate-dose enoxaparin (1 mg/kg Subcutaneously daily if BMI<30kg/m2 or 0.5 mg/kg Subcutaneously twice daily if BMI ≥ 30kg/m2).
  Other Names: intermediate dose Enoxaparin
  Arms: Interventional
Drug: Standard of Care thromboprophylaxis — Patients randomized to the standard of care arm will receive standard prophylactic dose enoxaparin (40 mg subcutaneously daily if BMI <30kg/m2 and 30 mg subcutaneously twice daily or 40 mg subcutaneously twice daily if BMI ≥ 30 kg/m2).
  Arms: Standard of Care

SUMMARY:
This prospective, randomized, open-label, multi-center interventional study is designed to compare the safety and efficacy of two LMWH dosing protocols in patients admitted to the University of Iowa Hospitals with COVID-19 who meet the modified ISTH Overt DIC criteria score ≥3. Patients will be randomized to standard prophylactic dose LMWH (standard of care arm) or intermediate-dose LMWH (intervention arm).

DETAILED DESCRIPTION:
Potentially eligible patients will be identified by a healthcare professional per institutional policy on privacy. The healthcare professional will assess the eligibility of the patient by performing a chart review which will include laboratory results and weight as measured on admission to the hospital. After obtaining verbal consent from the patient to be contacted for the study, a member of the research staff will approach the patient to be part of the study. The research staff will obtain informed consent from the patient/LAR before collecting any data and performing any procedures.

5.2 Trial interventions

As standard of care, hospitalized patients with confirmed COVID-19 will be monitored for coagulopathy. Daily blood tests for platelet count, prothrombin time, D-Dimer, and fibrinogen and weekly thromboelastography will be obtained, and a daily Modified ISTH Overt DIC score will be calculated (Exhibit 1). Only patients meeting all inclusion and exclusion criteria will be asked to participate in the trial. Patients will be randomized to one of two arms:

1. Patients randomized to the standard of care arm will receive standard prophylactic dose enoxaparin (40 mg subcutaneously daily if BMI <30 kg/m2; 30 mg subcutaneously twice daily or 40 mg subcutaneously twice daily if BMI ≥ 30 kg/m2).
2. Patients randomized to the intervention arm will receive intermediate-dose enoxaparin (1 mg/kg Subcutaneously daily if BMI <30 kg/m2 or 0.5 mg/kg Subcutaneously twice daily if BMI ≥ 30 kg/m2), with doses rounded up to the nearest dose syringe in hospitalized patients with laboratory confirmed SARS CoV-2 infection.

5.3 Dose Modifications

1. Enoxaparin will be held if platelets decrease to <25,000/mm3. Enoxaparin will resume once platelets increase to ≥25,000/ mm3.
2. Enoxaparin will be held if fibrinogen is <50 mg/dL. Enoxaparin will resume once fibrinogen increases to ≥50 mg/dL.
3. Enoxaparin will be held if estimated Creatinine clearance < 15 ml/min calculated by the modified Cockcroft and Gault formula and resumed once the Creatinine Clearance is ≥15 ml/min.
4. Enoxaparin will be held if there is a clinical suspicion for heparin induced thrombocytopenia.
5. Enoxaparin dose will be reduced by 25% if Creatinine Clearance ≥15 and <30 ml/min calculated by the modified Cockcroft and Gault formula and increased once the estimated Creatinine Clearance is ≥30 ml/min in both the arms.

All participating patients will continue the assigned doses of enoxaparin until hospital discharge or until a clinical event occurs requiring either discontinuation of anticoagulation therapy or full therapeutic dose anticoagulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmed SARS-CoV-2 infection
* Age ≥18 years
* Requires hospital admission for further clinical management
* Modified ISTH Overt DIC score ≥ 3

Exclusion Criteria:

* Indication for full therapeutic-dose anticoagulation
* Acute venous thromboembolism (deep vein thrombosis or pulmonary embolism) within prior 3 months
* Acute cardiovascular event within prior 3 months
* Acute stroke (ischemic or hemorrhagic) within prior 3 months
* Active major bleeding
* Severe thrombocytopenia (<25,000/mm3)
* Increased risk of bleeding, as assessed by the investigator
* Acute or chronic renal insufficiency with Creatinine Clearance < 30 ml/min calculated by the modified Cockcroft and Gault formula
* Weight < 40 kg
* Known allergies to ingredients contained in enoxaparin, allergy to heparin products or history of heparin induced thrombocytopenia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Gundersen Health System, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Tang N, Li D, Wang X, Sun Z. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 Apr;18(4):844-847. doi: 10.1111/jth.14768. Epub 2020 Mar 13. PMID 32073213
- [Background] Lentz SR. Thrombosis in the setting of obesity or inflammatory bowel disease. Hematology Am Soc Hematol Educ Program. 2016 Dec 2;2016(1):180-187. doi: 10.1182/asheducation-2016.1.180. PMID 27913478
- [Derived] Eustes AS, Palani Kumar MK, Peterson JA, Mast AE, Lentz SR, Dayal S. Elevated tissue factor pathway inhibitor delays thrombin generation in COVID-19 but is not associated with clinical outcomes. Blood Vessel Thromb Hemost. 2025 Apr 29;2(3):100071. doi: 10.1016/j.bvth.2025.100071. eCollection 2025 Aug. PMID 40765912
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Flumignan RL, Tinoco JDS, Pascoal PI, Areias LL, Cossi MS, Fernandes MI, Costa IK, Souza L, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Prophylactic anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD013739. doi: 10.1002/14651858.CD013739. PMID 33502773

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator: Standard of Care: Patients randomized to the standard of care arm will received standard prophylactic dose enoxaparin ( 40mg subcutaneously daily if BMI <30kg/m2 and 30 mg subcutaneously twice daily or 40 mg subcutaneously twice daily if BMI ≥ 30kg/m2).
- Other: Interventional: Patients randomized to the intervention arm will receive intermediate-dose enoxaparin (1 mg/kg Subcutaneously daily if BMI <30 kg/m2 or 0.5 mg/kg Subcutaneously twice daily if BMI ≥ 30kg/m2).
Period: Overall Study
Arm/Group | Active Comparator: Standard of Care | Other: Interventional
Started | 88 | 88
Completed | 85 | 84
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Did not receive assigned treatment | 1 | 3

BASELINE CHARACTERISTICS:
Population: From 88 starting in Standard of Care group, 2 withdrew prior to treatment leaving 86 remaining. From 88 starting in Interventional group, 1 withdrew prior to treatment leaving 87 remaining.
Groups:
- Standard of Care: Patients randomized to the standard of care arm will received standard prophylactic dose enoxaparin (40mg subcutaneously daily if BMI <30kg/m2 and 30 mg subcutaneously twice daily or 40 mg subcutaneously twice daily if BMI ≥ 30kg/m2).
- Interventional: Patients randomized to the intervention arm will receive intermediate-dose enoxaparin (1 mg/kg Subcutaneously daily if BMI <30 kg/m2 or 0.5 mg/kg Subcutaneously twice daily if BMI ≥ 30kg/m2).
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Interventional | Total
Number analyzed (Participants) | 86 | 87 | 173
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 42 | 89
  >=65 years | 39 | 45 | 84
Age, Continuous [Median (Full Range); unit: years] | 63.5 [30 to 85] | 65 [24 to 86] | 64 [24 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 40 | 76
  Male | 50 | 47 | 97
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 3 | 7 | 10
  Asian | 2 | 2 | 4
  Hispanic | 15 | 9 | 24
  White | 63 | 68 | 131
  Other | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 86 | 87 | 173
Median BMI - kg/m^2 [Median (Inter-Quartile Range); unit: kg/m^2] | 30.7 [27.2 to 35.8] | 30.0 [24.7 to 36.6] | 30.5 [25.9 to 36.2]
BMI ≥ 30 kg/m^2 [Count of Participants; unit: Participants] | 56 | 50 | 106
Time from COVID-19 test to enrollment [Median (Inter-Quartile Range); unit: Days] — Median time from positive COVID-19 test to enrollment - in days
  Days | 4.5 [1 to 9] | 5 [1 to 9] | 5 [1 to 9]
Coexisting Conditions [Number; unit: participants]
  Cancer | 13 | 7 | 20
  Diabetes mellitus | 34 | 30 | 64
  Heart Disease | 27 | 27 | 54
  Hypertension | 53 | 51 | 104
  Lung Disease | 19 | 20 | 39
  Obesity | 39 | 45 | 84
  Current or former smoker | 38 | 35 | 73
  Admitted to ICU | 54 | 53 | 107
Lab Value: D-dimer [Median (Inter-Quartile Range); unit: ng/mL fibrinogen equivalent units] | 1900 [870 to 3980] | 1570 [1030 to 4050] | 1680 [920 to 3980]
Lab Value: Prothrombin time [Median (Inter-Quartile Range); unit: seconds] | 11 [11 to 12] | 11 [11 to 12] | 11 [11 to 12]
Lab Value: Fibrinogen [Median (Inter-Quartile Range); unit: mg/dL] | 552 [461 to 654] | 543 [462 to 670] | 552 [461 to 666]
Lab Value: Platelet count [Median (Inter-Quartile Range); unit: 10^9 platelets/L] | 270 [204 to 358] | 257 [217 to 332] | 261 [207 to 358]
Lab Value: Absolute lymphocyte count [Median (Inter-Quartile Range); unit: 10^6 cells/L] | 735 [545 to 1460] | 800 [490 to 1230] | 781 [500 to 1310]
Other treatments for COVID-19 [Number; unit: participants] — Other treatments for COVID-19 in the intention-to-treat population during the trial period. The protocol allowed patients to receive other experiment or approved treatments for COVID-19.
  participants
    Azithromycin | 11 | 25 | 36
    Convalescent | 23 | 23 | 46
    Corticosteroids | 67 | 63 | 130
    Famotidine | 30 | 25 | 55
    Remdesivir | 54 | 51 | 105

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: All-cause mortality
Time Frame: 30 Days post intervention
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care: Patients randomized to the standard of care arm will received standard prophylactic dose enoxaparin ( 40mg subcutaneously daily if BMI <30kg/m2 and 30 mg subcutaneously twice daily or 40 mg subcutaneously twice daily if BMI ≥ 30kg/m2).
Arm/Group | Standard of Care | Interventional
Number analyzed (Participants) | 86 | 87
Participants | 18 | 13

2. Secondary Outcome: Number of Participants With Acute Kidney Injury
Description: Defined as an estimated creatinine clearance <30 mL/min
Time Frame: 30 days post intervention
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Interventional
Number analyzed (Participants) | 86 | 87
Participants | 15 | 11

3. Secondary Outcome: Number of Participants With Arterial Thrombosis
Description: Risk of ischemic stroke, myocardial infarction and/or limb ischemia
Time Frame: 30 Days post intervention
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Interventional
Number analyzed (Participants) | 86 | 87
Participants | 3 | 5

4. Secondary Outcome: Number of Participants With Venous Thrombosis
Description: Those at risk of symptomatic venous thromboembolism, which is a blood clot in a vein.
Time Frame: 30 Days post intervention
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Interventional
Number analyzed (Participants) | 86 | 87
Participants | 6 | 7

5. Secondary Outcome: Number of Participants With Major Bleeding
Description: Those at risk of ISTH defined major bleeding, such as fatal bleeding, or bleeding into a critical area or organ.
Time Frame: 30 Days post intervention
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Interventional
Number analyzed (Participants) | 86 | 87
Participants | 2 | 2

6. Secondary Outcome: Number of Participants With Minor Bleeding
Description: Defined as a bleeding event that did not meet ISTH criteria for major bleeding.
Time Frame: 30 Days post intervention
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Interventional
Number analyzed (Participants) | 86 | 87
Participants | 6 | 6

ADVERSE EVENTS:
Time Frame: 30 Days
Description: From 88 starting in Standard of Care group, 2 withdrew prior to treatment leaving 86 remaining. From 88 starting in Interventional group, 1 withdrew prior to treatment leaving 87 remaining.
Arm/Group | Standard of Care | Interventional
All-Cause Mortality (participants affected / at risk) | 18/86 | 13/87
Serious Adverse Events (participants affected / at risk) | 32/86 | 31/87
Other Adverse Events (participants affected / at risk) | 0/86 | 0/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=86) | Interventional (N=87)
Acute kidney injury (Renal and urinary disorders) | 15 | 11
Arterial thrombosis (Blood and lymphatic system disorders) | 3 | 5
Venous thrombosis (Blood and lymphatic system disorders) | 6 | 7
Major bleeding (Blood and lymphatic system disorders) | 2 | 2
Minor bleeding (Blood and lymphatic system disorders) | 6 | 6

LIMITATIONS AND CAVEATS:
The trial design was based on data available in early 2020 that suggested a mortality of up to 40% in hospitalized patients with severe COVID-19. Another limitation is that the results cannot be extrapolated to all patients hospitalized with COVID-19, because more than 85% of screened patients did not meet eligibility criteria. Lastly, this study was not designed to examine outcomes beyond 30 days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT04360824/Prot_SAP_000.pdf